CLINICAL TRIAL: NCT02042937
Title: Enhancing Gluteus Maximus Recruitment: a Randomized Controlled Pilot Trial
Brief Title: Enhancing Gluteus Maximus Recruitment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John H. Hollman, Ph.D., Associate Professor of Physical Therapy, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-009283
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Muscular Weakness
Keywords: Knee; Hip; Muscle Strength; Electromyography; Biomechanical Phenomena
MeSH Terms: conditions — Muscle Weakness | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No intervention
- Exercise (Experimental): Exercise to improve gluteus maximus recruitment
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise to improve gluteus maximus recruitment
  Arms: Exercise

SUMMARY:
Can participants enhance gluteus maximus recruitment during a single-leg squat test following a neuromuscular training program?

ELIGIBILITY:
Inclusion criteria

* female
* healthy, active individuals
* age 18-36
* walk without assistive device
* able to run, jump, squat without difficulty
* show evidence of hip muscle dysfunction on screening exam

Exclusion criteria

* history of knee ligament injury, knee surgery, patella dislocation
* knee pain traversing stairs, squatting or after prolonged sitting within 6 months of test
* joint line tenderness suggestive of meniscus pathology
* positive knee ligament stress tests

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Knee valgus angle | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Hollman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Hollman JH, Hohl JM, Kraft JL, Strauss JD, Traver KJ. Modulation of frontal-plane knee kinematics by hip-extensor strength and gluteus maximus recruitment during a jump-landing task in healthy women. J Sport Rehabil. 2013 Aug;22(3):184-90. doi: 10.1123/jsr.22.3.184. Epub 2013 Apr 9. PMID 23579368
- [Background] Hollman JH, Hohl JM, Kraft JL, Strauss JD, Traver KJ. Effects of hip extensor fatigue on lower extremity kinematics during a jump-landing task in women: a controlled laboratory study. Clin Biomech (Bristol). 2012 Nov;27(9):903-9. doi: 10.1016/j.clinbiomech.2012.07.004. Epub 2012 Jul 26. PMID 22840731
- [Background] Hollman JH, Ginos BE, Kozuchowski J, Vaughn AS, Krause DA, Youdas JW. Relationships between knee valgus, hip-muscle strength, and hip-muscle recruitment during a single-limb step-down. J Sport Rehabil. 2009 Feb;18(1):104-17. doi: 10.1123/jsr.18.1.104. PMID 19321910